CLINICAL TRIAL: NCT02579603
Title: A Twelve Week, Open-label, Randomised, Parallel-group Study Evaluating Safety, Tolerability and Pharmacokinetics (PK) of Oral Nintedanib in Combination With Oral Pirfenidone, Compared to Treatment With Nintedanib Alone, in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Safety, Tolerability and PK of Nintedanib in Combination With Pirfenidone in IPF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.222; 2015-000640-42 (EudraCT Number)
Expanded Access: Available
Record Dates: First submitted 2015-10-16; First posted 2015-10-19 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

ARMS (2):
- Nintedanib (Experimental): Nintedanib 150 mg bid
  Interventions: Drug: Nintedanib
- Nintedanib and Pirfenidone (Experimental): Nintedanib 150 mg bid combined with pirfenidone up to 801 mg tid
  Interventions: Drug: Nintedanib; Drug: Pirfenidone

INTERVENTIONS:
Drug: Nintedanib — Nintedanib 150mg bid
Drug: Pirfenidone
  Other Names: Pirfenidone 801 mg tid
  Arms: Nintedanib and Pirfenidone

SUMMARY:
This is a phase IV, twelve week, open label, randomized, parallel group study to assess safety and tolerability of combined treatment with nintedanib and pirfenidone.

A secondary objective is to assess the exposure based on PK trough concentration values to nintedanib either given alone or in combination with pirfenidone and to assess the exposure of pirfenidone when combined with nintedanib.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent consistent with ICH-GCP(The International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use- Good clinical practice) and local laws, signed prior to any study procedures being performed (including any required washout)
* Male or female patients aged greater than or equal to 40 years at visit 1
* Idiopathic Pulmonary Fibrosis (IPF) diagnosis, based upon the ATS (American Thoracic Society)/ERS (European Respiratory Society)/JRS (Japanese Respiratory Society)/ALAT (Latin American Thoracic Association) 2011 guideline and confirmed by the investigator based on chest high resolution computed tomography (HRCT) scan performed within 12 months of visit 1
* FVC (Forced vital capacity) greater than or equal to 50% of predicted normal at visit 1

Exclusion criteria:

* ALT (Alanine transaminase), AST (Aspartate aminotransferase)> 1.5 fold upper limit of normal (ULN) at visit 1
* Total bilirubin > 1.5 fold ULN at visit 1
* Relevant airways obstruction (i.e. pre-bronchodilator FEV1 (Forced Expiratory Volume in one second)/FVC <0.7) at visit 1
* History of myocardial infarction within 6 months of visit 1 or unstable angina within 1 month of visit 1
* Bleeding Risk: Known genetic predisposition to bleeding, Patients who require fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, dabigatran, heparin, hirudin etc) or high dose antiplatelet therapy, History of haemorrhagic central nervous system event within 12 months prior to visit 1, History of haemoptysis or haematuria, active gastro-intestinal bleeding or ulcers and/or major injury or surgery within 3 months prior to visit 1, International normalised ratio (INR) > 2 at visit 1, Prothrombin time and partial thromboplastin time (PTT) > 150% of institutional ULN at visit 1
* Planned major surgery during the trial participation, including lung transplantation,major abdominal or major intestinal surgery.
* History of thrombotic event (including stroke and transient ischemic attack) within 12 months of visit 1
* Severe renal impairment (Creatinine clearance <30 mL/min calculated by Cockcroft-Gault formula at visit 1) or end-stage renal disease requiring dialysis
* Treatment with NAC (n-acetylcysteine), prednisone >15 mg daily or >30 mg every 2 days OR equivalent dose of other oral corticosteroids and/or fluvoxamine within 2 weeks of visit 2
* Treatment with azathioprine, cyclophosphamide, cyclosporine as well as any other investigational drug within 8 weeks of visit 2
* Previous treatment with pirfenidone
* Permanent discontinuation of nintedanib in the past due to Adverse Events considered drug-related
* Known hypersensitivity to nintedanib, pirfenidone, peanut or soya or to any of the excipients
* A disease or condition which in the opinion of the investigator may interfere with testing procedures or put the patient at risk when participating in this trial
* Alcohol or drug abuse which in the opinion of the treating physician would interfere with treatment
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Women of childbearing potential not willing or able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly5 for 28 days prior to and 3 months after nintedanib administration
* Patients not able to understand and follow study procedures including completion of self administered questionnaires without help
* Patients who require dose reduction and/or temporary interruption during the run-in period with nintedanib 150 mg bid
* Patients with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-10-16 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (23):
- United States (6):
  - Western CT Medical Group, P.C., Danbury, Connecticut
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Minnesota Lung Center, Minneapolis, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Lowcountry Lung and Crit Care, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Concordia Hospital, Winnipeg, Manitoba
- France (7):
  - HOP Avicenne, Bobigny
  - HOP de la Cavale Blanche, Brest
  - HOP Louis Pradel, Bron
  - HOP Calmette, Lille
  - HOP Pasteur, Nice
  - HOP Bichat, Paris
  - HOP Pontchaillou, Rennes
- Germany (3):
  - Klinik Donaustauf, Donaustauf
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
- Italy (3):
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - Osp. S. Giuseppe Fatebenefratelli, Milan
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Netherlands (2):
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam

REFERENCES:
- [Derived] Vancheri C, Kreuter M, Richeldi L, Ryerson CJ, Valeyre D, Grutters JC, Wiebe S, Stansen W, Quaresma M, Stowasser S, Wuyts WA; INJOURNEY Trial Investigators. Nintedanib with Add-on Pirfenidone in Idiopathic Pulmonary Fibrosis. Results of the INJOURNEY Trial. Am J Respir Crit Care Med. 2018 Feb 1;197(3):356-363. doi: 10.1164/rccm.201706-1301OC. PMID 28889759

RESULTS

PARTICIPANT FLOW:
Groups:
- Nintedanib: Patients were orally administered Nintedanib 2x150 mg soft gelatine capsule daily (1 capsule of 150 mg twice daily) with the possibility to reduce to 2x100 mg daily (1 capsule of 100 mg twice daily).
- Nintedanib + Pirfenidone: Patients were orally administered Nintedanib 2x150 mg soft gelatine capsule daily (1 capsule of 150 mg twice daily) with the possibility to reduce to 2x100 mg daily (1 capsule of 100 mg twice daily) in combination with pirfenidone. The pirfenidone dose was titrated up to 2403 mg daily according to the following schedule: 801 mg (1 capsule of 267 mg 3 times daily) from Visit 3 until the phone call visit ; 1602 mg daily (2 capsules of each 267 mg 3 times daily) after the phone call visit; 2403 mg daily (3 capsules of each 267 mg 3 times daily) starting at Visit 4 after the PK sampling had been performed.The dose of pirfenidone could have been reduced to 1 or 2 capsule(s) 3 times daily.
Period: Overall Study
Arm/Group | Nintedanib | Nintedanib + Pirfenidone
Started | 52 (Started are the randomised patients) | 53 (Started are the randomised patients)
Number of Patients Treated | 51 | 53
Completed | 48 | 51
Not Completed | 4 | 2
Not completed — Not treated | 1 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Other than stated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set : The treated set (104 patients) consisted of all randomised patients who were dispensed study medication and were documented to have taken at least 1 dose of randomised investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib | Nintedanib + Pirfenidone | Total
Number analyzed (Participants) | 51 | 53 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.9 (6.8) | 68.9 (6.6) | 68.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 44 | 42 | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With On-treatment Gastrointestinal (GI) AEs (SOC GI Disorders) From Baseline to Week 12
Description: Percentage of patients with on-treatment gastrointestinal (GI) Adverse events (AEs) (SOC GI disorders) from baseline to week 12.
  On-treatment AEs were defined as AEs with an onset from the first dose of randomised treatment up to the last dose of randomised treatment (inclusive).
Time Frame: Baseline to week 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Nintedanib | Nintedanib + Pirfenidone
Number analyzed (Participants) | 51 | 53
percentage of participants | 52.9 | 69.8

2. Secondary Outcome: Predose Plasma Concentrations at Steady State (Cpre,ss) of Nintedanib at Baseline, Weeks 2 and 4
Description: Predose plasma concentrations at steady state (Cpre,ss) of nintedanib at baseline (Visit 3), Week 2 (Visit 4) and Week 4 (Visit 5)
Time Frame: baseline, prior to intake of study medication on week 2 and week 4
Population: Pharmacokinetic Set (PKS): This analysis set included all patients who had been treated with study medication and who provided evaluable data for at least 1 PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib | Nintedanib + Pirfenidone
Number analyzed (Participants) | 51 | 53
ng/mL
  baseline: number analyzed (Participants) | 46 | 46
  baseline | 7.08 (56.0) | 7.65 (72.5)
  Week 2: number analyzed (Participants) | 41 | 35
  Week 2 | 7.25 (52.7) | 8.17 (69.8)
  Week 4: number analyzed (Participants) | 44 | 30
  Week 4 | 5.92 (73.5) | 7.13 (63.9)

3. Secondary Outcome: Predose Plasma Concentrations at Steady State (Cpre,ss) of Pirfenidone
Description: Predose plasma concentrations at steady state (Cpre,ss) of pirfenidone at Week 2 (Visit 4) and Week 4 (Visit 5)
Time Frame: Prior to intake of study medication on week 2 and week 4
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib + Pirfenidone
Number analyzed (Participants) | 53
ng/mL
  Week 2: number analyzed (Participants) | 32
  Week 2 | 1120 (122)
  Week 4: number analyzed (Participants) | 28
  Week 4 | 1220 (90.7)

ADVERSE EVENTS:
Time Frame: From first dose administration of the study medication to 28 days after last drug administration; up to 124 days.
Description: Treated set was used. The treated set (104 patients) consisted of all randomised patients who were dispensed study medication and were documented to have taken at least 1 dose of randomised investigational treatment
Arm/Group | Nintedanib | Nintedanib + Pirfenidone
Serious Adverse Events (participants affected / at risk) | 5/51 | 2/53
Other Adverse Events (participants affected / at risk) | 36/51 | 46/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=51) | Nintedanib + Pirfenidone (N=53)
Atrial flutter (Cardiac disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=51) | Nintedanib + Pirfenidone (N=53)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 7
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 16 | 20
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 6 | 22
Vomiting (Gastrointestinal disorders) | 6 | 15
Asthenia (General disorders) | 3 | 1
Fatigue (General disorders) | 6 | 10
Pyrexia (General disorders) | 1 | 3
Hepatocellular injury (Hepatobiliary disorders) | 0 | 3
Bronchitis (Infections and infestations) | 2 | 5
Nasopharyngitis (Infections and infestations) | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 3
Weight decreased (Investigations) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Dizziness (Nervous system disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights